CLINICAL TRIAL: NCT02085811
Title: Screening for Kyphosis in the Mean Term in Patients Treated With Kyphoplasty Alone in the Management of Stable Traumatic Compression Fractures of the Thoracolumbar Spine
Acronym: KIPHO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: THOUANT-RICOLFI AOI 2012
Record Dates: First submitted 2014-03-05; First posted 2014-03-13 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2013-06

CONDITIONS: Thoracolumbar Spine
Keywords: Kyphoplasty; at a single level; (between T11 and L5); associated surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Patients
  Interventions: Other: radiography standard

INTERVENTIONS:
Other: radiography standard

SUMMARY:
The aim of this retrospective study is to show that kyphoplasty is a reliable technique in the treatment of certain traumatic vertebral fractures.

Patients will be selected from medical records archived at the Neuroradiology Department of Dijon CHU.

An information sheet and questionnaire will be sent to patients together with a letter to ask them to have a radiographic examination.

The radiographic images will be interpreted by two independent experts to evaluate the angle pf vertebral kyphosis.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged at least 18;
* who underwent Kyphoplasty between T11 and L5,
* Patients who had Kyphoplasty at a single level without associated surgery,
* Magerl type-A fracture.
* Non-tumoral and non-osteoporotic cause.

Exclusion Criteria:

* Compression fracture outside the T11-L5 segment, or fracture other than Magerl type A.
* Osteoporotic vertebral fracture
* Association with other post-traumatic fractures.
* History of Balloon Kyphoplasty, or of thoracic or lumbar spine surgery except simple discectomy.
* Pregnant or breast-feeding women
* Patients not covered by national health insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone kyphoplasty
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Measure of Spinal kyphosis angle | Between the post-operative period (D1) and a minimum of one year of follow-up

SECONDARY OUTCOMES:
Evaluation of pain (VAS) | At least 1 year after the kyphoplasty
Number of new vertebral fractures | At least 1 year after the kyphoplasty
Evaluation of quality of life (OSWESTRY and EIFEL) | At least 1 year after the kyphoplasty
Evolution of the regional angle of vertebral kyphosis | At least 1 year after the kyphoplasty

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de DIJON, Dijon, France